CLINICAL TRIAL: NCT05672524
Title: A Phase II Study of Induction Tucatinib and Trastuzumab With Total Neoadjuvant Therapy for Locally Advanced HER2-amplified Rectal Adenocarcinoma
Brief Title: A Study of Tucatinib and Trastuzumab in People With Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-185
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Adenocarcinoma of the Rectum; Locally Advanced Rectal Adenocarcinoma; Rectal Adenocarcinoma; HER2 Positive Rectal Adenocarcinoma; Rectal Cancer
Keywords: HER2 positive rectal adenocarcinoma; Adenocarcinoma; Adenocarcinoma of the Rectum; Locally Advanced Rectal Adenocarcinoma; Rectal Adenocarcinoma; Rectal Cancer; Tucatinib; Trastuzumab; Memorial Sloan Kettering Cancer Center; 22-185
MeSH Terms: conditions — Rectal Neoplasms; Adenocarcinoma | interventions — Trastuzumab; tucatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participant with Rectal Adenocarcinoma (Experimental): Participants will have HER2-positive locally advanced rectal adenocarcinoma.
  Interventions: Drug: Trastuzumab; Drug: Tucatinib

INTERVENTIONS:
Drug: Trastuzumab — Patients will then be given tucatinib (300 mg BID orally) and trastuzumab (8 mg/kg on day 1, then 6 mg/kg starting cycle 2 and every three weeks) therapy for an initial 6 week lead-in period. All patients, regardless of findings on rectal MRI will then transition to standard of care induction chemotherapy with continuation of the trastuzumab and tucatinib for a total of five additional cycles (15 extra weeks).
Drug: Tucatinib — Patients will then be given tucatinib (300 mg BID orally) and trastuzumab (8 mg/kg on day 1, then 6 mg/kg starting cycle 2 and every three weeks) therapy for an initial 6 week lead-in period. All patients, regardless of findings on rectal MRI will then transition to standard of care induction chemotherapy with continuation of the trastuzumab and tucatinib for a total of five additional cycles (15 extra weeks).

SUMMARY:
The study researchers believe that a combination of the drugs trastuzumab and tucatinib, given with standard chemotherapy (capecitabine and oxaliplatin/FOLFOX), may help participants with rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for the trial.
* Be ≥18 years of age on the date of signing informed consent.
* ECOG performance status of 0 or 1.
* Histologically confirmed rectal adenocarcinoma.
* Adenocarcinoma with distal margin of 15 cm or less from the anal verge on endoscopy, staged with endorectal ultrasound (ERUS) or magnetic resonance imaging (MRI) as cT3/cT4 N0 or cT(any) cN1/2,
* No evidence of distant metastases
* Radiologically measurable or clinically evaluable disease per Protocol Section 13.0.
* Have confirmed HER2-positive rectal adenocarcinoma, as defined by having tumor tissue tested at a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory, meeting at least one of the following criteria:

  1. HER2+ overexpression (3+ immunohistochemistry [IHC]) by an FDA-approved HER2 IHC test following the package insert's interpretational manual for gastric cancer
  2. HER2 2+ IHC is eligible if the tumor is amplified by an FDA-approved HER2 in situ hybridization assay (FISH or chromogenic in situ hybridization [CISH]) following the package insert's interpretational manual for gastric cancer
  3. HER2 (ERBB2) amplification by CLIA-certified Next Generation Sequencing (NGS) sequencing assay.
* Tumor specimen that demonstrates intact mismatch repair enzymes by immunohistochemistry or microsatellite stability as demonstrated by NGS or PCR.
* Tumor specimen that indicates RAS wild-type based on expanded RAS testing including KRAS exon 2 (codons 12 and 13), exon 3 (codons 59 and 61), and exon 4 (codons 117 and 146)
* Left ventricular ejection fraction >=50 assessed by echocardiography
* Negative pregnancy test done within 14 days prior to beginning treatment, for women of childbearing potential only. Subjects of childbearing potential must be willing to use an adequate method of contraception. Appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives, or double barrier method (diaphragm plus condom). Contraception is required for the course of the study starting with the first dose of study medication through 150 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Nonchildbearing potential is defined as follows (by other than medical reasons):

* ≥45 years of age and has not had menses for >1 year
* Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
* Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study.
* Demonstrate adequate organ function as defined in the Table 6-1 below within 14 days of Cycle 1 Day 1, all screening labs should be performed within 14 days of treatment initiation.

  * Absolute neutrophil count (ANC): ≥1,500 /mm3
  * Platelets: ≥100,000 / mcL
  * Hemoglobin: >9 g/dL or ≥5.6 mmol/L
  * Serum creatinine OR Measured or calculated creatinine clearance (Creatinine clearance should be calculated per institutional standard.) (GFR can also be used in place of creatinine or CrCl): ≤1.5 × upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 × institutional ULN
  * Serum total bilirubin: Total bilirubin ≤ 1.5 × upper limit of normal (ULN), except for subjects with known Gilbert's disease who may enroll if the conjugated bilirubin is ≥1.5 x ULN
  * AST (SGOT) and ALT (SGPT): ≤ 2.5 × ULN
  * International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT): For patients not taking warfarin: INR <1.5 or PT <1.5 x ULN; and either PTT or aPTT <1.5 x ULN. Patients on warfarin may be included on a stable dose with a therapeutic INR <3.5

Exclusion Criteria:

* Recurrent rectal cancer.
* Prior pelvic radiation therapy, chemotherapy, or surgery for rectal cancer.
* Tumor is causing symptomatic bowel obstruction (patients who have a temporary diverting ostomy are eligible).
* Other invasive malignancy ≤ 5 years prior to registration. Exceptions are non-melanoma skin cancer that has undergone potentially curative therapy and in situ cervical carcinoma.
* Active infection requiring systemic therapy.
* Other Anticancer or Experimental Therapy. No other experimental therapies (including chemotherapy, radiation, hormonal treatment, antibody therapy, immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, matrix metalloprotease inhibitors, thalidomide, anti-VEGF/Flk-1 monoclonal antibody or other experimental drugs) of any kind are permitted while the patient is receiving study treatment.
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
* Known active Hepatitis B (e.g., HbsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Any known chronic (non-transient) liver disease in the patient's past medical history such as (but not limited to) cirrhosis, NASH (non-alcoholic steatohepatitis) or NAFLD.
* Women who are pregnant or breastfeeding, or men expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening visit through 150 days after the last dose of study medication.
* Concurrent medical or psychiatric condition or disease which, in the investigator's judgement, would make them inappropriate candidates for entry into the study. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, chronic obstructive pulmonary disease, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
* Received a live vaccine within 30 days of planned start of study medication.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment.
* Inability to swallow pills or any significant gastrointestinal disease which would preclude the adequate oral absorption of medications
* Use of a strong cytochrome P450 (CYP)2C8 inhibitor that is not adequately cleared (five half-lives of elapsed time) before study initiation. In addition, use of a strong CYP3A4 or CYP2C8 inducer that is taken within 5 days prior to the first dose of study will also be an exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response of study participants | 21 +/- 4 weeks
  The primary objective of this trial is to determine the clinical complete response rate after the completion of initial neoadjuvant tucatinib and trastuzumab followed by standard of care induction chemotherapy (assessed around week 21 ± 4 weeks) in subjects with HER2-positive, RAS wild-type locally advanced rectal adenocarcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cercek, MD, Principal Investigator — Memorial Sloan Kettering Cancer
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center at Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org